CLINICAL TRIAL: NCT02889354
Title: Group-based Cognitive-behavioral Therapy for Adults With Attention-deficit/Hyperactivity Disorder Inattentive-type: a Pilot Study
Brief Title: Group-based Cognitive-behavioral Therapy for Adults With Attention-deficit/Hyperactivity Disorder Inattentive-type
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Benjamin Bohman, Principal Investigator, Karolinska Institutet
Allocation: Not Applicable | Model: Single Group | Purpose: Treatment
Other Study IDs: KI-2016/255-31/5
Record Dates: First submitted 2016-08-31; First posted 2016-09-05 (Estimated); Last update posted 2017-08-23 (Actual); Status verified 2017-08

CONDITIONS: Attention Deficit Disorder With Hyperactivity
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cognitive-behavioral therapy (Experimental)
  Interventions: Behavioral: Cognitive-behavioral therapy

INTERVENTIONS:
Behavioral: Cognitive-behavioral therapy

SUMMARY:
The newly developed CBT for ADHD inattentive-type (ADHD-I) protocol is tested for feasibility and acceptability in a pilot study with a single group design. The study also evaluates measurements and recruiting possibilities, and effects of the intervention. Research hypotheses include: 1. There is a basis for recruiting ADHD-I patients for participation in an RCT at psychiatric outpatient units, 2. The measurements in the study are feasible and reasonable in regards to patient characteristics; that is, the patients are responding to the questionnaires as intended, 3. The CBT for ADHD-I intervention is feasible in terms of treatment completion, compliance to home assignments, and credibility and relevance, and is lacking of or involves a tolerable degree of adverse effects, and 4. The CBT for ADHD-I protocol reduces core symptoms of ADHD-I as well as symptoms of stress, depression, and anxiety, and improves quality of life.

ELIGIBILITY:
Inclusion Criteria:

In addition to an ADHD inattentive-type diagnosis, inclusion criteria are:

1. 18 years or older,
2. intelligence quotient above 80-85, and
3. if on medication, it needs to be well-established since three months.

Exclusion Criteria:

1. autism spectrum disorder,
2. ongoing substance use disorder,
3. difficulties in compliance with medical or other treatment,
4. social and/or psychiatric problems to such an extent that it prevents focusing on treatment, or
5. ongoing cognitive-behavioral therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-08; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Brown ADD Scales | 14 weeks
  Diagnostic measure

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Bohman, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Capio Psykiatri AB, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No